CLINICAL TRIAL: NCT02859064
Title: A Phase II Study of Lanreotide in Patients With Metastatic Gastrointestinal Neuroendocrine Tumors Undergoing Liver-directed Radioembolization With Yttrium-90 Microspheres (SIR-Spheres®)
Brief Title: Study of Lanreotide in Patients With Metastatic Gastrointestinal Neuroendocrine Tumors Who Are Undergoing Liver-directed Radioembolization With Yttrium-90 Microspheres
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 221
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-07

CONDITIONS: Neuroendocrine Tumors; Gastrointestinal Neoplasms; Carcinoid Tumors
Keywords: radioembolization; somatostatin analogs; carcinoid; neuroendocrine; liver-directed therapy
MeSH Terms: conditions — Neuroendocrine Tumors; Gastrointestinal Neoplasms; Carcinoid Tumor | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lanreotide/Y-90 microspheres (Experimental): Lanreotide: 120 mg by subcutaneous injection (SQ) on Day 1 of every cycle (every 28 days) in combination with SIR-Spheres therapy.
  Y-90 (Yttrium-90) microspheres [SIR-Spheres therapy]: dose and treatment day to be determined by treating radiation oncologist.
  Interventions: Drug: Lanreotide; Device: Y-90 microspheres

INTERVENTIONS:
Drug: Lanreotide — Administered every 28 days irrespective of when SIR-Spheres is administered. No waiting or adjusting of schedule is required. Lanreotide treatment may continue monthly until disease progression or unacceptable toxicity occurs.
  Other Names: Somatuline® Depot Injection
Device: Y-90 microspheres — To be administered by injection through a trans-femoral catheter into the hepatic artery.
  Other Names: SIR-Spheres

SUMMARY:
Neuroendocrine tumors (NETs) and cancers that originate from the gastrointestinal tract can be resistant to standard chemotherapy and often metastasize to the liver. Lanreotide (Somatuline® Depot) Injection and Yttrium-90 microspheres (SIR-Spheres®) each have FDA approval to treat patients with metastatic NETs. The purpose of this study is to determine if treatment for patients with NETs can be optimized by combining these therapies.

DETAILED DESCRIPTION:
This is an open-label, prospective, multi-center Phase II study for patients with metastatic well-to-moderately differentiated neuroendocrine tumors, including typical carcinoid and pancreatic neuroendocrine tumors, who are candidates for liver-directed radioembolization.

Lanreotide (Somatuline® Depot) Injection, is FDA-approved for treating unresectable, well- or moderately-differentiated, locally advanced or metastatic gastroentero-pancreatic neuro-endocrine tumors (GEP-NETs) to improve progression-free survival. Radioembolization with yttrium-90 microspheres (SIR-Spheres® therapy) is FDA-approved for treating liver metastases from colorectal cancer. While each of these individual treatments has had promising results, investigators hypothesize that treatment for patients with NETs can be optimized by co-administration of both therapies. Patients will receive treatment with lanreotide (120 mg subcutaneously every 28 days) in combination with SIR-Spheres therapy. The dose and treatment day of SIR-Spheres will be determined by the treating radiation oncologist. Patients who are currently receiving or have previously received lanreotide are eligible, and treatment with lanreotide can continue monthly until disease progression or unacceptable toxicity. Up to 25 patients are planned for enrollment to be conducted at approximately 5 investigational sites in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic well-to-moderately differentiated (or low-grade) neuroendocrine carcinoma, including typical carcinoid or pancreatic islet cell carcinoma.
* Computerized tomography (CT) scan evidence of liver metastases which are not treatable by surgical resection or local ablation with curative intent at the time of study entry. If a CT scan is not possible, then an MRI may be used.
* Patients who are currently receiving or have previously received lanreotide or another somatostatin analogue are eligible. Previous treatment with lanreotide or another somatostatin analogue is not required for study entry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Adequate hematologic, hepatic and renal function.
* Male patients with female partners of childbearing potential and women patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 3 months (90 days) following last dose of study drug(s). Male patients must also refrain from donating sperm during their participation in the study and for 3 months after last dose of study drug(s).
* Life expectancy ≥ 3 months.
* Willingness and ability to comply with study and follow-up procedures.
* Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

* Anti-cancer therapy with the exception of lanreotide or another somatostatin analogue within 21 days or 5 half-lives (whichever is shorter) of starting study treatment.
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to Cycle 1 Day 1 or has not recovered from side effects of such therapy.
* Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
* Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks prior to study entry and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
* Clinically significant ascites, cirrhosis, portal hypertension, or thrombosis as determined by clinical or radiologic assessment.
* Pregnant or lactating.
* Acute or chronic liver, renal, or pancreas disease.
* Any of the following cardiac diseases currently or within the last 6 months:

  * Left Ventricular Ejection Fraction (LVEF) <45% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc interval >480 ms on screening electrocardiogram (ECG)
  * Unstable angina pectoris
  * Congestive heart failure (New York Heart Association (NYHA) ≥ Grade 2
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  * Valvular disease with significant compromise in cardiac function
* Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] greater than 180 mmHg or diastolic blood pressure (DBP) greater than100 mmHg) (patients with values above these levels must have their blood pressure (BP) controlled with medication prior to starting treatment).
* Currently receiving treatment with therapeutic doses of warfarin sodium. Low molecular weight heparin is allowed.
* Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Known diagnosis of human immunodeficiency virus, hepatitis B or hepatitis C. Lab test results will be confirmed by the treating physician prior to study enrollment using patient's records not more than 1 year old.
* Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Research Medical Center/HCA Midwest, Kansas City, Missouri
  - Tennessee Oncology PLLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanreotide/Y-90 Microspheres: Lanreotide: 120 mg by subcutaneous injection (SQ) on Day 1 of every cycle (every 28 days) in combination with SIR-Spheres therapy.
  Y-90 (Yttrium-90) microspheres [SIR-Spheres therapy]: dose and treatment day to be determined by treating radiation oncologist.
  Lanreotide: Administered every 28 days irrespective of when SIR-Spheres is administered. No waiting or adjusting of schedule is required. Lanreotide treatment may continue monthly until disease progression or unacceptable toxicity occurs.
  Y-90 microspheres: To be administered by injection through a trans-femoral catheter into the hepatic artery.
Period: Overall Study
Arm/Group | Lanreotide/Y-90 Microspheres
Started | 6
Completed | 0
Not Completed | 6
Not completed — Progressive Disease | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of treatment of lanreotide and Y-90 microspheres.
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: Treatment-emergent Adverse Events were assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Time Frame: From the day of the first dose to 30 days after the last dose of study medication, up to 52 months
Population: All enrolled patients who received at least one dose of both study medications, at least one dose of lanreotide and at least one dose of Y-90 microspheres.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Overall Response Rate
Description: Percentage of patients with confirmed complete or partial response (CR or PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1),: Complete Response (CR): Disappearance of all target and non-target lesions; Partial Response (PR): >=30% decrease in the sum of the diameters of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 12 weeks post-treatment with SIR-Spheres then every 8 weeks, up to 52 months
Population: All enrolled patients who received at least one full dose of lanreotide and y-90 microspheres
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
percentage of participants | 16.7

3. Secondary Outcome: Disease Control Rate
Description: Percentage of patients with CR, PR or stable disease (SD) according to RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1),: Complete Response (CR): Disappearance of all target and non-target lesions; Partial Response (PR): >=30% decrease in the sum of the diameters of target lesions; Stable Disease: Meeting neither criteria for PR or Progression (PD= greater than 20% increase in the sum of diameters of target lesions, or an unequivocal increase in a non-target lesion, or the appearance of new lesions). Disease Control Rate (DCR) = CR + PR + SD.
Time Frame: At 12 weeks post-treatment with SIR-Spheres then every 8 weeks, up to 52 months.
Population: All enrolled patients who received at least one full dose of lanreotide and y-90 microspheres.
Measure: Number; unit: percentage of participants
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
percentage of participants | 100

4. Secondary Outcome: Progression Free Survival
Description: The time from Day 1 of study drug administration to disease progression as defined by RECIST v1.1, or death on study. Per RECIST V1.1 criteria, progression is defined as a greater than 20% increase in the sum of diameters of target lesions, or an unequivocal increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 12 weeks post-treatment with SIR-Spheres then every 8 weeks, up to 52 months
Population: All enrolled patients who received at least one full dose of lanreotide and y-90 microspheres.
Measure: Median (Full Range); unit: months
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
months | 11 [3.6 to 51.4]

5. Secondary Outcome: Overall Survival
Description: The time from Day 1 of study drug administration until death from any cause.
Time Frame: At 12 weeks post-treatment with SIR-Spheres then every 8 weeks, up to 52 months
Population: All enrolled patients who received at least one full dose of lanreotide and y-90 microspheres.
Measure: Median (Full Range); unit: months
Arm/Group | Lanreotide/Y-90 Microspheres
Number analyzed (Participants) | 6
months | 11.5 [3.7 to 51.4]

ADVERSE EVENTS:
Time Frame: From the date of first dose to 30 days after last dose of study treatment, up to 52 months.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Arm/Group | Lanreotide/Y-90 Microspheres
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanreotide/Y-90 Microspheres (N=6)
Asthenia (Musculoskeletal and connective tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanreotide/Y-90 Microspheres (N=6)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Macular hole (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood lactic acid increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema annulare (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT02859064/Prot_SAP_000.pdf